CLINICAL TRIAL: NCT02347774
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Efficacy and Safety Trial of 12 Weeks of Treatment With Nebulized SUN-101 in Patients With COPD: GOLDEN-4 (Glycopyrrolate for Obstructive Lung Disease Via Electronic Nebulizer
Brief Title: Efficacy and Safety Trial of 12 Weeks of Treatment With Nebulized SUN-101 in Patients With COPD (GOLDEN-4)
Acronym: GOLDEN-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUN101-302
Record Dates: First submitted 2015-01-21; First posted 2015-01-27 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SUN-101 50 mcg BID eFlow (CS) nebulizer (Experimental): SUN-101 50 mcg Twice Daily (BID) via e-Flow (R) Closed System (CS) nebulizer
  Interventions: Drug: SUN-101 50 mcg BID eFlow (CS) nebulizer
- SUN-101 25 mcg BID e-Flow (CS) nebulizer (Experimental): SUN-101 25 mcg (BID) via e-Flow (R) Closed System (CS) nebulizer
  Interventions: Drug: SUN-101 25 mcg BID eFlow (CS) nebulizer
- Placebo BID Eflow (CS) nebulizer (Placebo Comparator): Placebo (BID) via e-Flow (R) Closed System (CS) nebulizer
  Interventions: Drug: Placebo eFlow (CS) nebulizer

INTERVENTIONS:
Drug: SUN-101 50 mcg BID eFlow (CS) nebulizer — SUN-101 50 mcg twice daily (BID) eFlow (R) Closed System (CS) nebulizer
  Arms: SUN-101 50 mcg BID eFlow (CS) nebulizer
Drug: SUN-101 25 mcg BID eFlow (CS) nebulizer — SUN-101 25 mcg BID eFlow (R) Closed System (CS) nebulizer
  Arms: SUN-101 25 mcg BID e-Flow (CS) nebulizer
Drug: Placebo eFlow (CS) nebulizer — Placebo BID eFlow (R) Closed System (CS) nebulizer
  Arms: Placebo BID Eflow (CS) nebulizer

SUMMARY:
This is a trial of 12 weeks of treatment with nebulized SUN-101 using an Investigational eFlow® Closed System (CS) nebulizer in subjects with chronic obstructive pulmonary disease (COPD) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD 2014) guidelines.

DETAILED DESCRIPTION:
This is a Phase 3, randomized, double-blind, placebo-controlled, parallel-group, multicenter, efficacy and safety trial of 12 weeks of treatment with nebulized SUN-101 using an Investigational eFlow® Closed System (CS) nebulizer in approximately 645 subjects with chronic obstructive pulmonary disease (COPD) according to the Global Initiative for Chronic Obstructive Lung Disease (GOLD 2014) guidelines.

SUN-101 or placebo will be administered twice daily as an oral inhalation using the investigational eFlow CS nebulizer.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients age ≥ 40 years, inclusive
2. A clinical diagnosis of COPD according to the GOLD 2014 guidelines
3. Current smokers or ex-smokers with at least 10 pack-year smoking history (eg, at least 1 pack/day for 10 years, or equivalent)
4. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1 < 80% of predicted normal and > 0.7 L during Screening (Visit 1)
5. Post-bronchodilator (following inhalation of ipratropium bromide) FEV1/FVC ratio < 0.70 during Screening (Visit 1)
6. Ability to perform reproducible spirometry according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines (2005)
7. Subject, if female ≤ 65 years of age and of child bearing potential, must have a negative serum pregnancy test at Visit 1. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study and must use an acceptable method of birth control: a) an oral contraceptive, an intrauterine device (IUD), implantable contraceptive, transdermal or injectable contraceptive for at least 1 month prior to entering the study with continued use throughout the study and for thirty days following participation; b) barrier method of contraception, eg, condom and /or diaphragm with spermicide while participating in the study; and/or c) abstinence
8. Willing and able to provide written informed consent
9. Willing and able to attend all study visits and adhere to all study assessments and procedures

Exclusion Criteria:

1. Severe comorbidities including unstable cardiac or pulmonary disease or any other medical conditions that would, in the opinion of the Investigator, preclude the subject from safely completing the required tests or the study, or is likely to result in disease progression that would require withdrawal of the subject
2. Concomitant clinically significant respiratory disease other than COPD (eg, asthma, tuberculosis, bronchiectasis or other non-specific pulmonary disease).
3. Recent history of COPD exacerbation requiring hospitalization or need for increased treatments for COPD within 6 weeks prior to Screening (Visit 1).
4. Use of daily oxygen therapy > 12 hours per day
5. Respiratory tract infection within 6 weeks prior to Screening (Visit 1)
6. Use of oral, intravenous, or intramuscular steroids within 3 months prior to Screening (Visit 1)
7. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma of the skin
8. Prolonged QTcF (> 450 msec for males and > 470 msec for females) during Screening (Visit 1) as determined from the report provided by the central laboratory, or history of long QT syndrome
9. History of or clinically significant on-going bladder outflow obstruction or history of catheterization for relief of bladder outflow obstruction within the previous 6 months
10. History of narrow angle glaucoma
11. History of hypersensitivity or intolerance to aerosol medications
12. Recent documented history (within the previous 3 months) of substance abuse
13. Significant psychiatric disease that would likely result in the subject not being able to complete the study, in the opinion of the Investigator
14. Participation in another investigational drug study where drug was received within 30 days prior to Screening (Visit 1) or current participation in another investigational drug trial, including a SUN-101 study
15. Previously received SUN-101 (active treatment; formerly known as EP-101)
16. Contraindicated for treatment with, or having a history of reactions/hypersensitivity to anticholinergic agents, beta2 agonists, or sympathomimetic amines

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 641 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sunovion Respiratory Development
Locations (45):
- United States (45):
  - SEC Lung, LLC, Andalusia, Alabama
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Pulmonary Associates, PA, Glendale, Arizona
  - Phoenix Medical Research Institute, LLC, Peoria, Arizona
  - Clinical Research Consortium, Tempe, Arizona
  - Center for Clinical Trials of Sacramento, Inc., Sacramento, California
  - Institute of HealthCare Assessment, Inc, San Diego, California
  - Innovative Clinical Research, Broomfield, Colorado
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Longmont Pulmonary and Critical Care, Longmont, Colorado
  - Ribo Research, LLC dba Peninsula Research Inc., Ormond Beach, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Pulmonary Care Research Group, PA, Winter Park, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Duluth Biomedical Research, LLC, Duluth, Georgia
  - Southeast Regional Research Group, Rincon, Georgia
  - Asthma and Allergy Center of Chicago, SC, River Forest, Illinois
  - LaPorte County Institute for Clinical Research, Michigan City, Indiana
  - George Stanley Walker, MD, New Orleans, Louisiana
  - Minnesota Lung Center, Minneapolis, Minnesota
  - CAR.E. Clinical Research, St Louis, Missouri
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Delaware Valley Clinical Research, Marlton, New Jersey
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - PharmQuest, Greensboro, North Carolina
  - Clinical Research of Lake Norman, Huntersville, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Southeastern Research Center, LLC, Winston-Salem, North Carolina
  - Liliestol Research LLC, Fargo, North Dakota
  - New Horizons Clinical Research, Cincinnati, Ohio
  - Remington-Davis, Inc, Columbus, Ohio
  - Sridhar Guduri, MD, Dublin, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Allergy Associates Research Center, Portland, Oregon
  - Lowcountry Lung and Critical Care, PA, Charleston, South Carolina
  - Easley Clinical Research, Easley, South Carolina
  - Gaffney Pharmaceutical Research, Gaffney, South Carolina
  - Spectrum Medical Research, LLC, Gaffney, South Carolina
  - Clinical Research of Charleston, Mt. Pleasant, South Carolina
  - CU Pharmaceutical Research, Rock Hill, South Carolina
  - Hope Clinical Research, Seneca, South Carolina
  - New Phase Research & Development, Knoxville, Tennessee
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Pulmonary Associates of Richmond, Inc, Richmond, Virginia
  - Multicare Pulmonary Specialists, Tacoma, Washington

REFERENCES:
- [Result] Kerwin E, Donohue JF, Goodin T, Tosiello R, Wheeler A, Ferguson GT. Efficacy and safety of glycopyrrolate/eFlow(R) CS (nebulized glycopyrrolate) in moderate-to-very-severe COPD: Results from the glycopyrrolate for obstructive lung disease via electronic nebulizer (GOLDEN) 3 and 4 randomized controlled trials. Respir Med. 2017 Nov;132:238-250. doi: 10.1016/j.rmed.2017.07.011. Epub 2017 Jul 19. PMID 28838685
- [Derived] Ohar J, Tosiello R, Goodin T, Sanjar S. Efficacy and safety of a novel, nebulized glycopyrrolate for the treatment of COPD: effect of baseline disease severity and age; pooled analysis of GOLDEN 3 and GOLDEN 4. Int J Chron Obstruct Pulmon Dis. 2018 Dec 18;14:27-37. doi: 10.2147/COPD.S184808. eCollection 2019. PMID 30587959
- [Derived] Ferguson GT, Kerwin EM, Donohue JF, Ganapathy V, Tosiello RL, Bollu VK, Rajagopalan K. Health-Related Quality of Life Improvements in Moderate to Very Severe Chronic Obstructive Pulmonary Disease Patients on Nebulized Glycopyrrolate: Evidence from the GOLDEN Studies. Chronic Obstr Pulm Dis. 2018 Jun 6;5(3):193-207. doi: 10.15326/jcopdf.5.3.2017.0178. PMID 30584583

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled were randomized. All subjects were to be followed for the full 12-week treatment period of the study, whether or not they continued on the study drug, .until the end of the treatment period.
  One subject randomized in error to the placebo arm was never dosed .
Period: Study Participation
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Started | 214 | 214 | 213 (One subject randomized in error to the placebo arm was never dosed .)
Completed | 199 | 193 | 188
Not Completed | 15 | 21 | 25
Not completed — Lost to Follow-up | 3 | 6 | 2
Not completed — Withdrawal by Subject | 8 | 9 | 15
Not completed — Adverse Event | 1 | 4 | 6
Not completed — withdrew consent | 1 | 1 | 1
Not completed — Met Prolonged QT criteria | 1 | 0 | 0
Not completed — non-compliance with study drug | 0 | 1 | 0
Not completed — incarceration | 1 | 0 | 0
Not completed — randomized in error | 0 | 0 | 1
Period: On Study Treatment
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Started | 214 | 214 | 213 (One subject randomized in error to the placebo arm was never dosed .)
Completed | 190 | 183 | 177
Not Completed | 24 | 31 | 36
Not completed — Adverse Event | 9 | 15 | 19
Not completed — Lack of Efficacy | 3 | 0 | 2
Not completed — non-complicance with study medication | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — withdrew consent | 9 | 8 | 12
Not completed — Lost to Follow-up | 2 | 6 | 1
Not completed — Met Prolonged QT criteria | 1 | 0 | 0
Not completed — ranomized in error | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: As noted in the participant flow section, One subject randomized in error to the placebo arm was never dosed .
Groups:
- Total: Total of all reporting groups
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer | Total
Number analyzed (Participants) | 214 | 214 | 212 | 640
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 119 | 109 | 111 | 339
  >=65 years | 95 | 105 | 101 | 301
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.20) | 63.6 (8.66) | 63.7 (9.26) | 63.3 (9.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 90 | 88 | 265
  Male | 127 | 124 | 124 | 375
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 3 | 8
  Not Hispanic or Latino | 211 | 212 | 209 | 632
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 26 | 27 | 19 | 72
  White | 188 | 185 | 192 | 565
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 214 | 214 | 212 | 640
Cardiovascular risk (low/high) and categories for high cardiovascular risk [Number; unit: participants]
  low cardiovascular risk | 80 | 78 | 76 | 234
  high cardiovascular risk | 134 | 136 | 136 | 406
  ischemic heart disease | 20 | 24 | 20 | 64
  cerebrovascular disease | 10 | 8 | 9 | 27
  peripheral arterial disease | 7 | 9 | 17 | 33
  clinically significant arrhythmia | 8 | 7 | 6 | 19
  heart failure | 4 | 4 | 6 | 14
  hypertension | 124 | 123 | 125 | 372
Background long-acting beta(2) agonist (LABA) use [Number; unit: participants]
  background LABA use = yes | 67 | 69 | 69 | 205
  background LABA use = no | 147 | 145 | 143 | 435
Forced expiratory volume in one second (FEV1) [Least Squares Mean (Standard Deviation); unit: liters] | 1.3506 (0.55380) | 1.3232 (0.50179) | 1.13355 (0.48612) | 1.3365 (0.51414)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) at Week 12
Description: All collected Spirometry was performed according to internationally accepted standards. Trough FEV1 at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose.
  All collected values were used in this analyses, regardless if the subject remained on randomized treatment or not, and regardless if the values might potentially be affected by other therapies or not Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: baseline and Week 12
Population: Intent to Treat (ITT) Population: all subjects who were randomized to treatment and received at least one dose of study medication. Subjects were analyzed based on the treatment they were randomized to.One subject randomized in error to the placebo arm was never dosed .
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
liters | 0.0847 (0.01423) | 0.0921 (0.01446) | 0.0111 (0.01452)
Statistical Analysis 1: Comparison: SUN-101 50 mcg BID eFlow (CS) Nebulizer vs Placebo BID Eflow (CS) Nebulizer; The change from baseline in trough FEV1 was analyzed using a mixed model repeated measures including terms for treatment, cardiovascular risk, background LABA use, visit week, visit week by treatment interaction, and baseline FEV1 as a covariate. An unstructured covariance matrix was used; Test type: Superiority — A sample size of 215 subjects per treatment would give ~ 90% power to detect a treatment difference of 80 mL in the change from baseline in trough FEV1 at Week 12 between each of the 2 SUN-101 dose groups and placebo at alpha= 0.05, assuming a standard deviation of 255 mL and using a 2-sided test; p = 0.0002, Least Mean Squared (SE); Least Mean Squared (SE) = 0.0736, 95% CI 2-sided [0.0346 to 0.1127], Standard Error of Mean 0.01989 — In order to control the family-wise Type I error rate, the Hochberg procedure (a tree-structured gatekeeping procedure) was used for comparisons of the primary efficacy endpoints and the key secondary efficacy endpoints
Statistical Analysis 2: Comparison: SUN-101 25 mcg BID e-Flow (CS) Nebulizer vs Placebo BID Eflow (CS) Nebulizer; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0001, Least Mean Squared (SE); Least Mean Squared (SE) = 0.0810, 95% CI 2-sided [0.0416 to 0.1204], Standard Error of Mean 0.02006 — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Change From Baseline in Trough Forced Expiratory Volume in 1 Second (FEV1) Week 12
Description: On-treatment Spirometry was performed according to internationally accepted standards. Trough FEV1 at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose.
  Only on-treatment values (which included only data collected while subjects were taking study drug) are used for this analysis. Values affected by other medication use were set to missing. Non-collected or missing data were not imputed for this analysis. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Week 12
Population: Intent to Treat (ITT) Population: all subjects who were randomized to treatment and received at least one dose of study medication. Subjects were analyzed based on the treatment they were randomized to.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
liters | 0.0890 (0.01479) | 0.0909 (0.01492) | 0.0069 (0.01502)
Statistical Analysis 1: Comparison: SUN-101 50 mcg BID eFlow (CS) Nebulizer vs Placebo BID Eflow (CS) Nebulizer; The change from baseline in trough FEV1 was analyzed using a mixed model repeated measures model including terms for treatment, cardiovascular risk, background LABA use, visit week, visit week by treatment interaction, and baseline FEV1 as a covariate. An unstructured covariance matrix was used; Test type: Superiority; p < 0.0001, Least Mean Squared (SE) — In order to control the family-wise Type I error rate, the Hochberg procedure (a tree-structured gatekeeping procedure) was used for comparisons of the primary efficacy endpoints and the key secondary efficacy endpoints; I; Least Mean Squared (SE) = 0.0820, 95% CI 2-sided [0.0417 to 0.1224], Standard Error of Mean 0.02055
Statistical Analysis 2: Comparison: SUN-101 25 mcg BID e-Flow (CS) Nebulizer vs Placebo BID Eflow (CS) Nebulizer; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.0001, Least Mean Squared (SE) — [p-value comment as in outcome 2, analysis 1]; Least Mean Squared (SE) = 0.0840, 95% CI 2-sided [0.0433 to 0.1246], Standard Error of Mean 0.02069

3. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC) at Week 12
Description: All collected Spirometry was performed according to internationally accepted standards. Trough FVC at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose.
  All collected values were used in the analyses, regardless if the subject remained on randomized treatment or not, and regardless if the values might potentially be affected by other therapies or not Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: baseline and Week 12
Population: Intent to Treat (ITT) Population: all subjects who were randomized to treatment and received at least one dose of study medication. Subjects were analyzed based on the treatment they were randomized to. One subject randomized in error to the placebo arm was never dosed .
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
liters | 0.1090 (0.02205) | 0.1346 (0.2239) | 0.0156 (0.02247)

4. Secondary Outcome: Change From Baseline in Trough Forced Vital Capacity (FVC)Week 12
Description: On-treatment Spirometry was performed according to internationally accepted standards. Trough FVC at Week 12 was defined as the mean of the values collected at two time points 30 minutes apart at approximately 24 hours (± 1 hour) after the previous morning dose.
  Only on-treatment values (which included only data collected while subjects were taking study drug) are used for this analysis. Values affected by other medication use were set to missing. Non-collected or missing data were not imputed for this analysis. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
liters | 0.1210 (0.02332) | 0.1385 (0.02354) | 0.0084 (0.02367)

5. Secondary Outcome: Change From Baseline in Health Status Measured by St. George's Respiratory Questionnaire (SGRQ) at Week 12/End of Study
Description: All collected Participants reported change in health status by using the SGRQ. The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD: symptoms, activity, and impacts. A score was calculated for each of these 3 subscales and a "Total" score was calculated. In each case the lowest possible value is 0 and the highest 100. Higher values correspond to greater impairment of health status.
  All collected values were used in the analyses, regardless if the subject remained on randomized treatment or not. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
units on a scale | -3.825 (0.8060) | -3.225 (0.8168) | -0.138 (0.8067)

6. Secondary Outcome: Change From Baseline in Health Status Measured by St. George's Respiratory Questionnaire (SGRQ) Week 12/End of Study
Description: On-treatment Participants reported change in health status by using the SGRQ. The SGRQ contains 50 items divided into 2 parts covering 3 aspects of health related to COPD: symptoms, activity, and impacts. A score was calculated for each of these 3 subscales and a "Total" score was calculated. In each case the lowest possible value is 0 and the highest 100. Higher values correspond to greater impairment of health status.
  Only on-treatment values (which included only data collected while subjects were taking study drug) are used for this analysis. Values affected by other medication use were set to missing. Non-collected or missing data were not imputed for this analysis. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
units on a scale | -3.609 (0.8237) | -3.637 (0.8269) | -0.052 (0.8212)

7. Secondary Outcome: Change in Number of Rescue Medication Puffs Per Day Over the 12-week Double-blind Treatment Period
Description: All collected Participants completed an electronic diary (eDiary) daily (night time) to record the number of puffs of rescue medication inhaled in the previous 24 hours. A negative change from baseline indicates improvement.
  All collected values were used in the analyses, regardless if the subject remained on randomized treatment or not. Values not collected remained as missing values and were assumed to be missing at random (MAR).
Time Frame: Week 0-12
Population: Intent to Treat (ITT) Population: all subjects who were randomized to treatment and received at least one dose of study One subject randomized in error to the placebo arm was never dosed .
  medication. Subjects were analyzed based on the treatment they were randomized to.One subject randomized in error to the placebo arm was never dosed .
Measure: Least Squares Mean (Standard Error); unit: puffs (medication used)
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
puffs (medication used) | -0.845 (0.1311) | -0.959 (0.1310) | -0.678 (0.1339)

8. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAE)
Description: On-treatment A TEAE is defined as any non-serious AE that occurred on or after the first dose of study medication and within 7 days after the last dose of study medication, or any serious AE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent AE is an on-treatment AE.
Time Frame: Week 0-12
Population: Safety population was defined as all subjects who were randomized to treatment and received at least one dose of study medication.One subject randomized in error to the placebo arm was never dosed .
Measure: Count of Participants; unit: Participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
Participants | 114 | 101 | 111

9. Secondary Outcome: Percentage of Subjects With Treatment Emergent Adverse Events (TEAE)
Description: A TEAE is defined as any non-serious AE that occurred on or after the first dose of study medication and within 7 days after the last dose of study medication, or any serious AE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent AE is an on-treatment AE.
Time Frame: Week 0-12
Population: Safety population was defined as all subjects who were randomized to treatment and received at least one dose of study medication. One subject randomized in error to the placebo arm was never dosed .
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
percentage of participants | 53.3 | 47.2 | 52.4

10. Secondary Outcome: Number of Subjects With Treatment Emergent Serious Adverse Events (SAE)
Description: A treatment emergent SAE is defined as any SAE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent SAE is an on-treatment SAE.
Time Frame: Week 0-12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
Participants | 8 | 5 | 13

11. Secondary Outcome: Percentage of Subjects With Treatment Emergent Serious Adverse Events (SAE)
Description: as for outcome 10
Time Frame: Week 0-12
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
percentage of participants | 3.7 | 2.3 | 6.1

12. Secondary Outcome: Number of Subjects Who Discontinue Treatment Due to TEAE
Description: A TEAE is defined as any AE that occurred on or after the first dose of study medication and within 7 days after the last dose of study medication, or any serious AE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent AE is an on-treatment AE.
Time Frame: Week 0-12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
Participants | 9 | 15 | 19

13. Secondary Outcome: Percentage of Subjects Who Discontinue Treatment Due to TEAE
Description: as for outcome 12
Time Frame: Week 0-12
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
percentage of participants | 4.2 | 7.0 | 9.0

14. Secondary Outcome: Number of Subjects With Major Adverse Cardiac Events (MACE)
Description: All deaths and any other findings suggestive of a potential MACE (including clinically relevant information and SAEs, and all PTs form the SMQs "myocardial infarction", "other ischemic heart disease", "central nervous system hemorrhages and cerebrovascular conditions") were sent to an adjudication committee for review and categorized as CV death, nonfatal MI, and nonfatal stroke. The MACE score was defined as the total number of subjects with CV deaths, nonfatal MIs, and nonfatal strokes. These events were collected for the double-blind period (from the first date of study medication until the date of last contact)
Time Frame: Week 0-12
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
Participants
  MACE score | 0 | 0 | 0
  cardiovascular death | 0 | 0 | 0
  non-fatal myocardial infarction | 0 | 0 | 0
  non-fatal stroke | 0 | 0 | 0

15. Secondary Outcome: Percentage of Subjects With Major Adverse Cardiac Events (MACE)
Description: as for outcome 14
Time Frame: Week 0-12
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
percentage of participants
  MACE score | 0 | 0 | 0.9
  cardiovascular death | 0 | 0 | 0
  non-fatal myocardialinfarction | 0 | 0 | 0.9
  non-fatal stroke | 0 | 0 | 0

16. Secondary Outcome: Incidence Rate Per 1000 Person-years of Subjects With Major Adverse Cardiac Events (MACE)
Description: All deaths and any other findings suggestive of a potential MACE (including clinically relevant information and SAEs, and all PTs form the SMQs "myocardial infarction", "other ischemic heart disease", "central nervous system hemorrhages and cerebrovascular conditions") were sent to an adjudication committee for review and categorized as CV death, nonfatal MI, and nonfatal stroke. The MACE score was defined as the total number of subjects with CV deaths, nonfatal MIs, and nonfatal strokes. These events were collected for the double-blind period (from the first date of study medication until the date of last contact)
  Incidence rate: TT= Total Time in years. Total Time (TT) is defined as the time from the first date of study drug until the latter of the date of last contact or 30 days after the date of last dose. Incidence Rate (per 1000 person-years) = n/TT x 1000.
Time Frame: Week 0-12
Population: as for outcome 8
Measure: Number; unit: incidence rate
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Number analyzed (Participants) | 214 | 214 | 212
incidence rate | 64.6 | 63.0 | 62.2

ADVERSE EVENTS:
Time Frame: Week 0-12
Description: A treatment emergent SAE is defined as any SAE that occurred on or after the first dose of study medication and within 30 days after the last dose of study medication. A treatment emergent SAE is an on-treatment SAE.
Arm/Group | SUN-101 50 mcg BID eFlow (CS) Nebulizer | SUN-101 25 mcg BID e-Flow (CS) Nebulizer | Placebo BID Eflow (CS) Nebulizer
Serious Adverse Events (participants affected / at risk) | 8/214 | 5/214 | 13/212
Other Adverse Events (participants affected / at risk) | 41/214 | 47/214 | 39/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUN-101 50 mcg BID eFlow (CS) Nebulizer (N=214) | SUN-101 25 mcg BID e-Flow (CS) Nebulizer (N=214) | Placebo BID Eflow (CS) Nebulizer (N=212)
haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
artiral fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
artiral flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
cardiomyoathy (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
pancreatitis necrotising (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 3 (4)
chest injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
coronary artery restenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1)
nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SUN-101 50 mcg BID eFlow (CS) Nebulizer (N=214) | SUN-101 25 mcg BID e-Flow (CS) Nebulizer (N=214) | Placebo BID Eflow (CS) Nebulizer (N=212)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 17 (17) | 17 (19)
cough (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 14 (14) | 14 (14)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 16 (16) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study , the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.